CLINICAL TRIAL: NCT02842723
Title: Phase II Study on the Management of Pediatric Craniopharyngioma by a Combination of Partial Surgical Resection, and Protontherapy
Brief Title: Management of Pediatric Craniopharyngioma by a Combination of Partial Surgical Resection, and Protontherapy (Craniopharyngioma)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2008-01
Record Dates: First submitted 2016-07-11; First posted 2016-07-25 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Craniopharyngioma
Keywords: craniopharyngioma; protontherapy
MeSH Terms: conditions — Craniopharyngioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Protontherapy (Experimental)
  Interventions: Radiation: Protontherapy

INTERVENTIONS:
Radiation: Protontherapy — 59,5 Gy (1,7 Gy daily, 5 fractions per week).

SUMMARY:
Prospective, open labelled, phase II, monocenter trial to combine partial surgery resection and protontherapy to management paediatric craniopharyngioma.

DETAILED DESCRIPTION:
This study is phase II prospective, open labelled, phase ii, monocenter. The main objective is to evaluate the fractionated high precision radiotherapy with a dose of 59,5 Gy (1,7 Gy daily, 5 fractions per week).

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented craniopharyngioma
* Age range between 3 and 16 years
* Landsky performance status > 60
* Incomplete surgical resection or simple biopsy
* Solid and/or cystic aspect on imaging
* Irradiation performed at the time of presentation or of local progression
* Signed informed consent by parents or by legal representative (with copy to each participating center)

Exclusion Criteria:

* Previous history of radiotherapy (including stereotactic) administered to the head and neck region
* Severe vasculopathy
* Participation to a concurrent study
* Contra-indication to general anesthesia in children below 5 years
* Patient non-compliant to a minimum 30 mn immobilisation
* Patient deprived of freedom or under guardianship
* Patient not expected to be followed in a long run

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
local control rate at 3 years of a minimally aggressive surgical resection, followed by fractionated high precision radiotherapy | at 3 years

SECONDARY OUTCOMES:
visual pathway tolerance according to NCI-CTC v3.0 scale | through study completion, up to 9 years

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut Curie, Paris
  - Groupe Hospitalier Necker Enfants Malades, Paris
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA